CLINICAL TRIAL: NCT02322034
Title: Effects of Interval Training on Hormonal Pathways in Chronic Heart Failure
Brief Title: Interval Training and Hormones in Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Francesco Giallauria, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNINA-34/13
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; multiple neurohormonal axis disequilibrium; growth hormone deficiency; Insulin-like growth factor-1 (IGF-1); metabolic deficiency syndrome; interval training
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interval Training (Experimental): Hospital outpatient-based regimen (3 times/week for 24 weeks) exercise program will be performed by cycling for 4 minutes with 1-minute rest between intervals. High intensity exercise will be 90-95% peak heart rate. The exercise intensity will be established, and maintained throughout the 24-week exercise training period, by calculating the heart rate range as a percentage of maximum (90-95%) as obtained from the most recent cardiopulmonary exercise test. Every 4 weeks during the training program, the exercise intensity will be titrated to the same relative percentage of maximum (90-95%) as it is assumed most patients will become fitter over the training period.
  Interventions: Other: Interval Training
- Controls (No Intervention): CHF patients allocated to the control group (no intervention) will undergo biochemical and hormonal sampling, Doppler-echocardiography, cardiopulmonary exercise stress testing at study enrollment and at 24-week follow-up.

INTERVENTIONS:
Other: Interval Training — Exercise training protocol (high intensity, interval training) is followed by the enrolled patients on hospital outpatient-based regimen 3 times/week for 24 weeks. The high intensity group will perform interval cycling for 4 minutes with 1-minute rest between intervals. High intensity exercise will be 90-95% peak heart rate. The exercise intensity will be established, and maintained throughout the 24-week exercise training period, by calculating the heart rate range as a percentage of maximum (90-95%) as obtained from the most recent cardiopulmonary exercise test. Every 4 weeks during the training program, the exercise intensity will be titrated to the same relative percentage of maximum (90-95%) as it is assumed most patients will become fitter over the training period.
  Other Names: High Intensity Training; Intermittent Training
  Arms: Interval Training

SUMMARY:
The investigators aim at investigating whether 24-week high intensity interval training might exert beneficial effects by modulating neurohormonal axis in patients with chronic heart failure (CHF). Furthermore, the effect of detraining on neurohormonal axis in CHF patients will be evaluated.

DETAILED DESCRIPTION:
According to European Society of Cardiology the prevalence of Heart Failure (HF) is between 2 and 3% in general population and increases with age, so the prevalence in 70- to 80-years-old people is between 10 and 20%. HF is the cause of 5% of acute hospital admissions, is present in 10% of patients in hospital beds, and accounts for high national expenditure on health, mostly due to the cost of hospital admissions. Although some patients can live for many years and the great improvement of medical therapy during last decades, overall 50% of patients are dead at 4 years.

Despite different hypothesis that explain the underlying physiopathology of heart failure have been proposed over time, no single paradigm for heart failure was established definitively. One logical explanation of the inability to define the syndrome of heart failure in precise mechanistic model is that the clinical syndrome of heart failure almost certainly represents the summation of multiple anatomic, functional, and biological alterations that interact together in a complex way. Thus, it is not surprising that investigators have used a variety of complex model in an attempt to describe the syndrome of heart failure. Nowadays, the most accepted hypothesis explaining HF physiopathology and its progression is the "neurohormonal model". According to this paradigm, heart failure progresses as a result of the overexpression of biologically active molecules that exert toxic effects on the heart and circulation. A variety of molecules including norepinephrine, angiotensin II, endothelin, aldosterone, and tumor necrosis factor have been implicated as some of the factors that contribute to disease progression in the failing heart.

Despite the effectiveness of the neurohormonal model to explain disease progression and the many insights that it provided for the development of new therapies, there is increasing clinical evidence that suggests that our current models fail to completely explain disease progression. Thus, neurohormonal models may be necessary but not sufficient to explain all aspects of disease progression in the failing heart.

Because the prognosis of HF patients is still unsatisfactory despite optimal therapies, other mechanisms that contribute to HF progression need to be elucidated. Mounting evidence suggest that in heart failure there is a metabolic imbalance characterized by a predominance of the catabolic status over anabolic drive. The most impressive example is seen in end-stage HF known as "cardiac cachexia" characterized by strong weight loss, particularly lean mass and rapid deterioration of clinical conditions, attributed to a prevalence of catabolic pathways. If the hormonal imbalance is an epiphenomenon or an important pathophysiological mechanism in the HF progression is still matter of debate.

In particular deficit of each anabolic axis (adrenal, gonadal and somatotropic axes) is an independent marker of poor prognosis in HF patients and the coexistence of more than one deficiency identifies a subgroup of patients with a higher mortality.

The most involved hormonal axes include growth hormone (GH), its tissue effector insulin-like growth factor-1 (IGF-1), thyroid hormone, and anabolic steroids. Taken together, these alterations could be recognized as a multiple hormonal and metabolic deficiency syndrome (MHD) in HF patients. MHD has a significant impact on cardiac performance and HF progression.

The most involved hormonal axes include growth hormone (GH), its tissue effector insulin-like growth factor-1 (IGF-1), thyroid hormone, and anabolic steroids. Taken together, these alterations could be recognized as a multiple hormonal and metabolic deficiency syndrome (MHD) in HF patients. MHD has a significant impact on cardiac performance and HF progression.

Moreover, a pattern of Insulin-resistance (IR) is quite common in diabetic as well as non-diabetic CHF patients. IR has been found in about 30% of non-diabetic CHF patients and was related to underlying disease severity. Few studies have considered reduction of IR as a new therapeutic target.

In brief, it could be argued that CHF patients showed an anabolic/catabolic imbalance due to multiple neurohormonal axis disequilibrium. Anabolic hormonal deficiency is usually described in men with chronic heart failure (CHF) contributing to the anabolic/catabolic imbalance ultimately resulting in skeletal muscle waist and cardiac cachexia. Counteracting the anabolic deficit seems to play beneficial clinical effects in CHF patients. In fact, the increase of serum levels of testosterone and growth hormone (GH)/insulin-like growth factor 1 (IGF-1) axis obtained by hexogen administration, improves key symptoms of CHF such as exercise intolerance and muscle fatigue and positively impact quality of life. Besides the hexogen administration, an increase of the levels of anabolic hormones can be obtained through physical exercise. In healthy subjects, testosterone may increase remarkably as an acute response to both endurance and heavy resistance exercise. Similarly, GH concentrations generally increase in response to both strength and endurance exercise thereby stimulating IGF-1 production. Although this hormonal modulation could be one of the mechanisms by which exercise training exerts its beneficial effects on CHF patients, there are few data on endogenous exercise-induced increase of anabolic hormones in such patients.

Aside from the nature of the training activity, the effects of training may vary with different dose parameters, specifically program length, session duration and frequency and workload or intensity. In the most severely impaired patients, with initial exercise intolerance, sessions may initially be limited to 3-5 minutes duration with 3 or 4 sessions completed during the course of the day; however, recent work has suggested that if total exercise energy expenditure is standardized then intermittent exercise training programs may elicit superior benefits to heart failure patients compared to continuous exercise training sessions.

High intensity, repeated intermittent work periods separated by recovery periods have been shown to be efficacious in heart failure patients, and interval stress has been shown to be as effective as continuous workloads in older, healthy and post coronary artery bypass surgery populations. In a systematic review of 81 heart failure ExT studies only two of these reported peak VO2 changes of 10% and 20% respectively compared with 16.5% overall change in continuous exercise training and similar improvements with strength training. The underlying theory is that higher intensity, intermittent stress is more likely to promote peripheral adaptations and produce concurrent improvements in functional capacity. Recent work has shown that reductions of brain natriuretic peptide, a marker of myocardial stretch, may be greater in high intensity (90% peak VO2), rather than moderate intensity (70% peak VO2) exercise training in patients with severe left ventricular dysfunction. A recent meta-analysis showed that intermittent exercise elicits superior improvements in peak VO2 and VE/VCO2 slope compared to continuous exercise training in heart failure patients.

Few studies evaluated the hormonal response to interval training in CHF. However, the relatively small sample size, the lack of control group or the relatively short time exercise intervention limits the conclusions.

The present study aims at investigating whether 24-week high intensity interval training might exert beneficial effects by modulating neurohormonal axis in CHF patients. Furthermore, the effect of detraining on neurohormonal axis in CHF patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Stable New York Heart Association (NYHA) class II or III
* Resting left ventricular ejection fraction below 40%
* Measured peak VO2 below 14 ml/kg/min [Patients must be stable on prescribed cardiac medication for 1 month prior to entering the study]

Exclusion Criteria:

* myocardial infarction within 12 months prior to study entry;
* unstable angina; resting systolic blood pressure above 200 mmHg, or diastolic blood pressure above 110 mmHg;
* fever of unknown significance;
* critical aortic stenosis (peak systolic pressure gradient > 50 mm Hg with an aortic valve orifice area < 0.75 cm2 in average size adult);
* uncontrolled atrial or ventricular arrhythmias such as uncontrolled sinus tachycardia (> 120 beats.min-1);
* II or greater atrio-ventricular block;
* active pericarditis or myocarditis;
* recent embolism and thrombophlebitis;
* uncontrolled diabetes HbA1C%>9.5%;
* severe orthopedic or other medical conditions that would prohibit exercise;
* metabolic conditions such as acute thyroiditis, hypokalemia or hyperkalemia and hypovolemia;
* severe renal dysfunction (i.e. creatinine plasma levels >2.5 mg/dl);
* severe concomitant non-cardiac diseases such as cancer, dementia or any systemic disease limiting exercise;
* inability to participate in a prospective study for any logistic reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
peak exercise oxygen consumption (VO2peak) | 24 weeks
  cardiopulmonary functional capacity

SECONDARY OUTCOMES:
growth hormone (GH) - insulin-like growth factor-1 (IGF-1) | 24-week
  GH/IGF-1 axis balance
brain natriuretic peptide | 24-week
  BNP assay

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Vigorito, MD, Study Director — Federico II University of Naples
Locations (1):
- Division of Internal Medicine and Cardiac Rehabilitation, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arcopinto M, Isgaard J, Marra AM, Formisano P, Bossone E, Vriz O, Vigorito C, Sacca L, Douglas PS, Cittadini A. IGF-1 predicts survival in chronic heart failure. Insights from the T.O.S.CA. (Trattamento Ormonale Nello Scompenso CArdiaco) registry. Int J Cardiol. 2014 Oct 20;176(3):1006-8. doi: 10.1016/j.ijcard.2014.07.003. Epub 2014 Jul 11. No abstract available. PMID 25037691
- [Background] Isgaard J, Arcopinto M, Karason K, Cittadini A. GH and the cardiovascular system: an update on a topic at heart. Endocrine. 2015 Feb;48(1):25-35. doi: 10.1007/s12020-014-0327-6. Epub 2014 Jun 28. PMID 24972804
- [Background] Cittadini A, Marra AM, Arcopinto M, Bobbio E, Salzano A, Sirico D, Napoli R, Colao A, Longobardi S, Baliga RR, Bossone E, Sacca L. Growth hormone replacement delays the progression of chronic heart failure combined with growth hormone deficiency: an extension of a randomized controlled single-blind study. JACC Heart Fail. 2013 Aug;1(4):325-330. doi: 10.1016/j.jchf.2013.04.003. Epub 2013 Aug 5. PMID 24621936
- [Background] Smart NA, Dieberg G, Giallauria F. Intermittent versus continuous exercise training in chronic heart failure: a meta-analysis. Int J Cardiol. 2013 Jun 20;166(2):352-8. doi: 10.1016/j.ijcard.2011.10.075. Epub 2011 Nov 17. PMID 22100179
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the diagnosis and treatment of acute and chronic heart failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur J Heart Fail. 2008 Oct;10(10):933-89. doi: 10.1016/j.ejheart.2008.08.005. Epub 2008 Sep 16. No abstract available. PMID 18826876
- [Background] Mann DL. Mechanisms and models in heart failure: A combinatorial approach. Circulation. 1999 Aug 31;100(9):999-1008. doi: 10.1161/01.cir.100.9.999. No abstract available. PMID 10468532
- [Background] Jankowska EA, Biel B, Majda J, Szklarska A, Lopuszanska M, Medras M, Anker SD, Banasiak W, Poole-Wilson PA, Ponikowski P. Anabolic deficiency in men with chronic heart failure: prevalence and detrimental impact on survival. Circulation. 2006 Oct 24;114(17):1829-37. doi: 10.1161/CIRCULATIONAHA.106.649426. Epub 2006 Oct 9. PMID 17030678
- [Background] Doehner W, Rauchhaus M, Ponikowski P, Godsland IF, von Haehling S, Okonko DO, Leyva F, Proudler AJ, Coats AJ, Anker SD. Impaired insulin sensitivity as an independent risk factor for mortality in patients with stable chronic heart failure. J Am Coll Cardiol. 2005 Sep 20;46(6):1019-26. doi: 10.1016/j.jacc.2005.02.093. PMID 16168285
- [Background] Taegtmeyer H. Cardiac metabolism as a target for the treatment of heart failure. Circulation. 2004 Aug 24;110(8):894-6. doi: 10.1161/01.CIR.0000139340.88769.D5. No abstract available. PMID 15326079
- [Background] Anker SD, Chua TP, Ponikowski P, Harrington D, Swan JW, Kox WJ, Poole-Wilson PA, Coats AJ. Hormonal changes and catabolic/anabolic imbalance in chronic heart failure and their importance for cardiac cachexia. Circulation. 1997 Jul 15;96(2):526-34. doi: 10.1161/01.cir.96.2.526. PMID 9244221
- [Background] Caminiti G, Volterrani M, Iellamo F, Marazzi G, Massaro R, Miceli M, Mammi C, Piepoli M, Fini M, Rosano GM. Effect of long-acting testosterone treatment on functional exercise capacity, skeletal muscle performance, insulin resistance, and baroreflex sensitivity in elderly patients with chronic heart failure a double-blind, placebo-controlled, randomized study. J Am Coll Cardiol. 2009 Sep 1;54(10):919-27. doi: 10.1016/j.jacc.2009.04.078. PMID 19712802
- [Background] Iellamo F, Manzi V, Caminiti G, Vitale C, Castagna C, Massaro M, Franchini A, Rosano G, Volterrani M. Matched dose interval and continuous exercise training induce similar cardiorespiratory and metabolic adaptations in patients with heart failure. Int J Cardiol. 2013 Sep 10;167(6):2561-5. doi: 10.1016/j.ijcard.2012.06.057. Epub 2012 Jul 4. PMID 22769574
- [Background] Caminiti G, Iellamo F, Manzi V, Fossati C, Cioffi V, Punzo N, Murugesan J, Volterrani M, Rosano G. Anabolic hormonal response to different exercise training intensities in men with chronic heart failure. Int J Cardiol. 2014 Oct 20;176(3):1433-4. doi: 10.1016/j.ijcard.2014.08.040. Epub 2014 Aug 13. No abstract available. PMID 25150472